CLINICAL TRIAL: NCT04970134
Title: Spanish Observational Study for MOLecular Characterization of THYroid Carcinoma MOLTHY Project
Brief Title: Spanish Study for Molecular Characterization of Thyroid Carcinoma
Acronym: MOLTHY
Status: Active, not recruiting | Type: Observational
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Responsible Party: Sponsor
Other Study IDs: TTCC-2020-02
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Differentiated Thyroid Carcinoma; Medullary Thyroid Carcinoma
Keywords: advanced and/or metastatic disease; iodine refractory
MeSH Terms: conditions — Carcinoma, Medullary | interventions — Immunohistochemistry; In Situ Hybridization, Fluorescence; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tumor sample from each patient in formalin-fixed paraffin block (FFPE)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thyroid carcinoma: Advanced and / or metastatic thyroid carcinoma with initial histological diagnosis date before January 1, 2021 of the types:
  Differentiated thyroid carcinoma (DTC) refractory to radio-iodine, including papillary carcinomas, follicular carcinomas, poorly differentiated carcinomas of the thyroid and the different corresponding variants.
  Medullary thyroid carcinoma (MTC).
  Interventions: Other: Immunohistochemistry (IHC); Other: Fluorescence In-Situ Hybridization (FISH); Other: Oncomine Focus Assay Platform with 52 genes

INTERVENTIONS:
Other: Immunohistochemistry (IHC) — VENTANA pan-TRK technique (EPR17341) Assay, with Optiview DAB-detection kit and Optiview amplification kit. Using FFPE slices
Other: Fluorescence In-Situ Hybridization (FISH) — FISH using FFPE slices for genes: Neurotrophic tyrosin kinase 1 (NTRK1), Neurotrophic tyrosin kinase 3 (NTRK3) and rearranged during transfection (RET)
Other: Oncomine Focus Assay Platform with 52 genes — Oncomine Focus Assay Platform with 52 genes (35 Hotspot genes, 19 Copy number variants and 23 Gene fusions). Using FFPE slices
  Other Names: Next Generation Sequencing (NGS)

SUMMARY:
This project is a retrospective observational study based on the molecular characterization of a Spanish population of patients with refractory radio-iodine differentiated thyroid cancer (DTC) and medullary thyroid carcinoma (MTC) with advanced and / or metastatic disease undergoing systemic treatment, or under clinical observation.

Three diagnostic techniques will be performed on formalin-fixed paraffin embedded (FFPE) tumor samples from the study population: immunohistochemistry (IHC), fluorescence by in situ hybridization (FISH) as well as Next-Generation Sequencing (NGS) techniques by means of DNA and RNA analysis (Ion Platform Torrent - Oncomine Focus Assay, 52 gene detection). The results of each patient will be compared in order to correlate the results of each method.

DETAILED DESCRIPTION:
Immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH) techniques will be carried out to identify NTRK and RET alterations. NTRK alterations will be identified using IHC techniques (NTRK over-expression), and FISH techniques (break-apart method). RET alterations will also be identified using the FISH technique (break-apart method).

At the same time, DNA and RNA will be extracted for sequencing techniques using the Oncomine Focus Assay platform, including 52 genes (35 Hotspot genes, 19 Copy number variants and 23 Gene fusions, including NTRK and RET).

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be over 18 years old
2. Obtaining the informed consent signed by the patient or his legal representative.
3. Have a paraffinized tumor sample available for analysis in the central laboratory, preferably from total thyroidectomy.
4. Life expectancy greater than 6 months.
5. Thyroid carcinoma with a date of initial histological diagnosis before January 1, 2021 of the types:

(1) Differentiated thyroid carcinoma (DTC) refractory to radio-iodine, including papillary carcinomas, follicular carcinomas, poorly differentiated thyroid carcinomas, and the corresponding different variants. The radio-refractoriness criteria will be defined by medical criteria and / or by decision of the tumor committee (depending on the organization of each hospital) or (2) Medullary thyroid carcinoma (MTC). 6. Potential candidate patients must meet at least one of the following premises:

1. Patients with advanced / metastatic disease in wait & see follow-up.
2. Patients with advanced / metastatic disease currently undergoing treatment or in progression to any type of multikinase inhibitor, such as, for example: sorafenib, lenvatinib, cabozantinib, axitinib, vandetanib, ...
3. Patients with advanced / metastatic disease under treatment or in progression to treatments that inhibit immune checkpoints (anti programed death (PD-1) or its ligand (PD-L1), anti Cytotoxic T-Lymphocyte Antigen 4 (CTLA-4), others) or who are participating in clinical trial regimen. They must be patients who have previously progressed to multikinase inhibitors.

Exclusion Criteria:

1. Patients affected by other malignant histologies not mentioned in the previous section (eg melanoma, lymphoma, sarcoma, ...) or benign tumors exclusively of the thyroid gland.
2. Patients with radioiodine sensitive differentiated thyroid carcinoma or anaplastic thyroid carcinomas.
3. Patients with refractory radioiodine differentiated thyroid carcinoma and advanced medullary thyroid carcinomas with the possibility of local ablative treatment with radical or curative intent (surgery, radiosurgery, radio-ablation, ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated to include 150 patients over 18 years of age with thyroid carcinoma (radioiodine resistant differentiated thyroid carcinoma and medullary thyroid carcinoma) undergoing systemic treatment or under clinical follow-up.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Throughout the study. Approximately 2 years
  Time from start of data capture (retrospectively) to progression disease. Patients may be stratified in subgroups attending to their histologic subtype and molecular genetic profile.
Overall survival (OS) | Throughout the study. Approximately 2 years
  Time from start of data capture (retrospectively) to death. Patients may be stratified in subgroups attending to their histologic subtype and molecular genetic profile.
Objective response rate | Throughout the study. Approximately 2 years
  Response to systemic treatments received if available. Patients may be stratified in subgroups attending to their histologic subtype and molecular genetic profile.
Prevalence of genetic alterations | Throughout the study. Approximately 2 years
  Frequency of genetic alterations in the study population determined by the molecular genetic interventions: IHC, FISH and NGS

CONTACTS AND LOCATIONS:
Overall Officials: Neus Basté Rotllan, M.D. Ph.D., Principal Investigator — Hospital Clinic of Barcelona
Locations (12):
- Spain (12):
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Durán i Reinals, L'Hospitalet de Llobregat, Barcelona
  - Fundació Althaia, Manresa, Barcelona
  - Consorci Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital universitario Marqués de Valdecilla, Santander, Cantabria
  - Institut Català d'Oncologia Girona - ICO Girona, Girona, Girona
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza